CLINICAL TRIAL: NCT04116762
Title: Does the Use of TissuePAtchDS-P Allow for Day Case PArotid Surgery? A Randomised Controlled Superiority Trial Comparing TissuePatchDS-P Versus Surgical Drain in Benign Superficial Parotidectomy.
Brief Title: TissuePAtchDS--P ™ PArotidectomy Trial.
Acronym: TAPAS
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: All 3 participants receiving intervention in assessment phase developed seromas
Sponsor: Poole Hospital NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SP170310A
Record Dates: First submitted 2019-10-03; First posted 2019-10-07 (Actual); Last update posted 2019-10-16 (Actual); Status verified 2019-10

CONDITIONS: Parotid Gland Disorders

STUDY DESIGN:
Intervention Model Description: 1. The first part is to perform a pilot study at the lead site only, which will recruit 5 patients to have their surgery using TissuePatchDS-P alone to ensure that the product is safe to use and that no immediate complications are observed.
  2. If the pilot data suggests that TissuePatch is not associated with immediate, short or medium term complications (as confirmed by the investigators, sponsor and independent Trial Steering Committee) the trial will progress to the randomised controlled phase. A total of 50 patients will be recruited from the outpatient setting at participating National Health Service (NHS) trusts - 25 will be randomised to the control group (surgical drain) and 25 will be randomised to the intervention arm (TissuePatch).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Placement of TissuePatchDS-P™ at time of operation. No surgical drain is used.
  Interventions: Device: TissuePatchDS-P™
- Control (Active Comparator): No use of TissuePatchDS-P™. Wound is closed with a surgical drain (Surgeon's choice) in situ.
  Interventions: Device: Surgical Drain

INTERVENTIONS:
Device: TissuePatchDS-P™ — The therapy to be used in the intervention arm is TissuePatchDS-P™. This is a preformed, standard-sized artificial adhesive that will be used between the parotid tissue and subcutaneous tissue. It can be cut to an appropriate size for the defect. The intention of this installation is to seal and close the potential space that is created with removal of superficial parotid tissue
  Arms: Intervention
Device: Surgical Drain — A surgical drain used in superficial parotid surgery is a thin polyvinylchloride (PVC) tube, with perforations at the end, which is placed at the end of the procedure before the surgical wound is closed in the cavity created following removal of parotid tissue. The tube is connected to a closed vacuum system attached to a plastic bottle outside of the patient's body which acts to remove the fluid that collects after an operation.
  Arms: Control

SUMMARY:
The parotid (salivary) gland can develop growths (tumours), most of which are not cancerous but may develop into a cancer if left untreated. Tumours located near the surface of the gland are surgically removed in a procedure called a superficial parotidectomy. Post-surgery, fluid accumulates in the space left behind by the gland and currently, this is managed via insertion of a surgical drain (tube attached to a vacuumed bottle). Patients are then routinely admitted to hospital for 24-48 hours until it is safe for the drain to be removed.

As well as the need for a prolonged hospital stay, there are known risks associated with drains e.g. infection, fluid collection under the skin (seroma) and communication between parotid tissue and the skin (fistula). This study aims to evaluate the effectiveness of applying an adhesive sealant (TissuePatchDS-P) between the parotid gland and the skin after removal of a non-cancerous parotid tumour. This would be instead of a surgical drain, as the sealant closes the space and should prevent fluid build-up. This may allow for same-day discharge and reduce complications.

DETAILED DESCRIPTION:
The parotid (salivary) gland can develop growths (tumours), most of which are not cancerous but may develop into a cancer if left untreated. Tumours located near the surface of the gland are surgically removed in a procedure called a superficial parotidectomy. Post-surgery, fluid accumulates in the space left behind by the gland and currently, this is managed via insertion of a surgical drain (tube attached to a vacuumed bottle). Patients are then routinely admitted to hospital for 24-48 hours until it is safe for the drain to be removed.

As well as the need for a prolonged hospital stay, there are known risks associated with drains e.g. infection, fluid collection under the skin (seroma) and communication between parotid tissue and the skin (fistula). This study aims to evaluate the effectiveness of applying an adhesive sealant (TissuePatchDS-P) between the parotid gland and the skin after removal of a non-cancerous parotid tumour. This would be instead of a surgical drain, as the sealant closes the space and should prevent fluid build-up. This may allow for same-day discharge and reduce complications.

As no trials to date have used TissuePatchDS-P without a surgical drain, this study will run in two phases - an assessment/pilot phase with 5 participants using TissuePatchDS-P only. This will include compulsory overnight stay and ultrasound scan within 24 hours to ensure safety before progressing to the randomised controlled trial phase. In this phase, 50 participants will be randomised to receive either: surgical drain (standard care) or TissuePatchDS-P. After surgery, patients in both groups will be reviewed by their care team and discharged when appropriate.

Participants will be followed up at their routine 6-week post-surgical visit and then a trial doctor will conduct a study-related telephone consultation at 3 months post-surgery for long-term assessment of safety, clinical outcomes and quality of life.

ELIGIBILITY:
Inclusion Criteria:

1. All patients undergoing superficial parotidectomy for benign parotid disease.
2. Patients 18 years of age or above.

Exclusion Criteria:

1. American Society of Anesthesiologists (ASA) classification >2 and/or Body Mass Index (BMI) >35.
2. Any patient with malignant, infected/inflamed or recurrent parotid disease.
3. Patients taking immunosuppressants.
4. Patients with a history of allergic reaction to the composites of the patch
5. Previous parotid surgery to the same side.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2018-11-30 (Actual); Primary Completion 2019-10-01 (Actual); Study Completion 2019-10-01 (Actual)

PRIMARY OUTCOMES:
Proportion of participants discharged at day 0 following superficial parotidectomy. | Day one

SECONDARY OUTCOMES:
Number of complications | Three months
  Number of complications (e.g. haematoma, seroma, salivary fistula and symptomatic Frey's syndrome)
European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire Head and Neck Module (EORTC QLQ-HN35) | Three months

CONTACTS AND LOCATIONS:
Locations (1):
- Poole Hospital NHSFT, Poole, Dorset, United Kingdom

IPD SHARING:
Plan to Share IPD: No